CLINICAL TRIAL: NCT01799239
Title: Investigating the Safety and Performance of Newly Developed 1-piece Ostomy Product Concept Compared With SenSura 1-piece in Subjects With an Ileostomy
Brief Title: Safety and Performance of Newly Developed 1-piece Ostomy Product Compared With SenSura
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CP237
Record Dates: First submitted 2013-02-22; First posted 2013-02-26 (Estimated); Results first posted 2013-12-05 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-08

CONDITIONS: Ileostomy - Stoma
Keywords: stoma ileostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- First Test product; then SenSura (Experimental): The subject in this arm first test the Test product The test product is a newly developed ostomy appliance with a new top film. Due to company confidentiality the product is not described in further details.
  After cross-over the subject test SenSura which is CE-marked and commerical available.
  Interventions: Device: Test product; Device: SenSura
- First SenSura, Then Test product (Active Comparator): The subject in this arm first test SenSura which is CE-marked and commerical available.
  After cross-over the subject test the Test product The test product is a newly developed ostomy appliance with a new top film. Due to company confidentiality the product is not described in further details.
  Interventions: Device: Test product; Device: SenSura

INTERVENTIONS:
Device: Test product — The test product consists of an adhesive with a new top film
Device: SenSura — SenSura is the CE-marked and commercially available comparator product

SUMMARY:
The aim of the current investigation is to evaluate the combination of an adhesive with a soft top film.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Be able to handle the bags themselves
4. Have an ileostomy with a diameter between 15 and 55 mm
5. Have had their ileostomy for at least 3 months
6. Currently use a 1-piece flat ostomy appliance with open bag
7. Use minimum 1 product every second day, i.e. maximum 2 days wear time
8. Be suitable for participation in the study and for using a standard adhesive, flat base plate
9. Must be able and willing to use custom cut products
10. Accept to test two 1-piece products within the study period

Exclusion Criteria:

1. Use irrigation during the study period (flush the intestines with water)
2. Currently receiving or have within the past 2 months received chemotherapy or radiation therapy
3. Currently receiving or have within the past month received systematic steroid or local treatment in the peristomal area
4. Are pregnant or breastfeeding
5. Participating in other interventional clinical investigations or have previously participated in this investigation
6. Currently using a ostomy belt
7. Currently using extended wear product
8. Have a loop ileostomy
9. Known hypersensitivity towards any of the test products
10. Suffering from severe peristomal skin problems prior to participation in the investigation (assessed by the study nurse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Carter, MSc, Study Chair — Coloplast A/S
Locations (1):
- Skövde Hospital, Skövde, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were recruited from hospital sites in Sweden and in Germany subjects were recruit from the Coloplast database and from hospital sites.
Pre-assignment Details: The investigation was designed as a cross-over study where subjects that did not complete the 1 period as planned were allowed to continue to the next test period.
Groups:
- First Test Product; Then SenSura: The subjects tested two products: In the first period the subjects tested the newly developed ostomy bag called Test product. In the second period the subjects tested the comparator SenSura
- First SenSura, Then Test Product: The subjects tested two products: In the first period the subjects tested the comparator SenSura. In the second period the subjects tested the newly developed ostomy bag called Test product
Period: Period 1 (7 Days)
Arm/Group | First Test Product; Then SenSura | First SenSura, Then Test Product
Started | 15 (It was uncertain in which order the product were tested for 1 subject. Subject is excl from analysis) | 16 (It was uncertain in which order the product were tested for 1 subject. Subject is excl from analysis)
Completed | 12 | 15
Not Completed | 3 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Protocol Violation | 0 | 1
Period: Period 2 (7 Days)
Arm/Group | First Test Product; Then SenSura | First SenSura, Then Test Product
Started | 13 | 15
Completed | 11 | 14
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Three subjects were excluded from the intention to treat (ITT) population. Two of the were inclusion criteria violaters; 1 convex user and 1 colostomist. with the last subject it was uncertain in which order the subject tested the test products. the subejct was excluded from the analysis
Groups:
- Overall Study: Describing baseline data for all subjects in the ITT population
Arm/Group | Overall Study
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Leakage (Percentage of All Baseplates With Leakage)
Description: leakage is measured using a 4-point leakage scale developed by Coloplast A/S. At every baseplate change the subjects had to look at the skin facing side of the baseplate and access which of the four scenarios described below provided an accurate description of the baseplate.
  The subjects tick of one of the four possible answers:
  1. No leakage
  2. Starting to leak (leakage under the baseplate)
  3. Leakage (seepage of faeces resulting in leakage on clothes)
  4. Sudden leakage (the baseplate pops off resulting in sudden leakage under the baseplate and outside the baseplate)
Time Frame: After each baseplate change over a period, of 7 days
Measure: Number; unit: percentage baseplates with leakage
Units Other Than Participants: Baseplates
Groups:
- Test Product: The new test product is a 1-piece open ostomy product with the intended use being collecting output from an ileostomy.
- SenSura: CE marked and launched SenSura used in this investigation is a 1-piece open appliance with the intended use being to collect output from an ileostomy.
Arm/Group | Test Product | SenSura
Number analyzed (Participants) | 29 | 26
Number analyzed (Baseplates) | 184 | 167
percentage baseplates with leakage | 34 | 35

ADVERSE EVENTS:
Time Frame: The adverse events were collected for 14 days
Description: The subject for whom it was unknown which intervention was recieved did not have any adverse events in the course of the study
Arm/Group | Test Product | SenSura
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 1/32 | 1/32
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product (N=32) | SenSura (N=32)
pain in the peristomal area (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Itching in the peristomal area (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
red skin in the peristomal area (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less